CLINICAL TRIAL: NCT00689078
Title: Single Center, Randomized, Double-Masked Evaluation of the Efficacy of PredAcetate 1% Ophthalmic Suspension Compared to Pred Acetate 0.12% Ophthalmic Suspension, Lot Etab 0.2% Ophthalmic Suspension, and Placebo in a Modified CAC Model
Brief Title: Evaluation of the Efficacy of Topical Ophthalmic Steroids in a Modified Conjunctival Allergen Challenge (CAC) Model
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-003-05
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — prednisolone acetate; Methylprednisolone; Loteprednol Etabonate; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pred acetate 1% (Active Comparator): Prednisolone acetate 1.0% in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Interventions: Drug: Prednisolone Acetate 1%
- Pred acetate .12% (Active Comparator): Prednisolone acetate 0.12% in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Interventions: Drug: Prednisolone Acetate 0.12%
- Lot Etab 0.2% (Active Comparator): Loteprednol Etabonate 0.2% in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Interventions: Drug: Loteprednol Etabonate 0.2%
- Placebo (Placebo Comparator): Tears Naturale (Artificial Tears) in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone Acetate 1% — One drop in both eyes (OU) BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Other Names: Pred Forte (Allergan)
  Arms: Pred acetate 1%
Drug: Prednisolone Acetate 0.12% — One drop in both eyes (OU) BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Other Names: Pred Mild (Allergan)
  Arms: Pred acetate .12%
Drug: Loteprednol Etabonate 0.2% — One drop in both eyes (OU) BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Other Names: Alrex (Bausch & Lomb)
  Arms: Lot Etab 0.2%
Drug: Placebo — One drop in both eyes (OU) BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
  Other Names: Tears Naturale; Artificial tears
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of prednisolone acetate 1% ophthalmic suspension as compared to prednisolone acetate 0.12% ophthalmic suspension, loteprednol etabonate 0.2% ophthalmic suspension, and placebo (Tears Naturale® II) in the prevention of the signs and symptoms of allergic conjunctivitis. Comparisons will be made following 1 week of twice daily (BID) dosing and 1 week of four times daily (QID) dosing.

DETAILED DESCRIPTION:
Structure:

Prospective, single center, randomized, double-masked, parallel treatment comparison study. Subjects will be randomized to one of the following treatment arms to be dosed bilaterally twice daily (BID) for the first dosing period and four times daily (QID) for the second dosing period:

1. Prednisolone Acetate 1% ophthalmic suspension
2. Prednisolone Acetate 0.12% ophthalmic suspension
3. Loteprednol Etabonate 0.2% ophthalmic suspension
4. Tears Naturale® II

Duration:

Approximately four (4) weeks

Controls:

Artificial Tears (Tears Naturale® II)

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age & either sex, any race
* Willing and able to follow all instructions
* Positive history of ocular allergies
* Reproducible positive ocular allergic reaction induced by conjunctival allergen challenge

Exclusion Criteria:

* Have planned surgery during trial period
* Female currently pregnant, planning a pregnancy or lactating
* Use of disallowed medications
* Have ocular infections, or ocular conditions that could affect study parameters
* Have moderate to severe dry eye
* Have used an investigational drug or device within 30 days of start of study
* Female that is currently pregnant, planning a pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Torkildsen, MD, Principal Investigator — American board of Ophthalmology
Locations (1):
- Ophthalmic Research Associates, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one site in the US.
Pre-assignment Details: Participant flow and baseline characteristics are presented for the 36 subjects that met all inclusion and none of the exclusion criteria and were randomized to receive Pred Forte, Pred Mild, Alrex, or Tears Naturale. 36 subjects were enrolled, 4 discontinued, and 32 subjects completed the study.
Groups:
- Pred Forte; Pred Mild; Alrex; Tears Naturale: 1 drop in each eye up to 4 times daily for up to 4 weeks
Period: Overall Study
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Started | 9 | 9 | 9 | 9
Intent to Treat | 9 | 7 | 8 | 8
Completed | 9 | 7 | 8 | 8
Not Completed | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Pred Forte: Prednisolone acetate 1.0% in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
- Pred Mild: Prednisolone acetate 0.12% in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
- Alrex: Loteprednol Etabonate 0.2% in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
- Tears Naturale (Placebo): Tears Naturale (Artificial Tears) in each eye BID starting at Visit 2 (Day 0) for 6 days. Then in each eye QID starting the day after Visit 5 (Day 21) for 6 days.
- Total: Total of all reporting groups
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale (Placebo) | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.11 (6.15) | 44.11 (11.53) | 44.67 (18.65) | 45.78 (14.71) | 43.67 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 3 | 16
  Male | 5 | 5 | 4 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching at Baseline (Day 0)
Description: A baseline CAC was performed on Day 0. Post-CAC ocular itching from Day 0 will be compared to post-CAC ocular itching, post-instillation, on Day 6, Day 7, Day 27 and Day 28. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 9 | 9 | 9
units on a scale
  3 minutes post-CAC | 2.53 (0.507) | 3.08 (0.771) | 2.61 (0.953) | 2.5 (0.781)
  5 minutes post-CAC | 2.92 (0.661) | 3.47 (0.475) | 3.06 (0.682) | 2.75 (0.612)
  7 minutes post-CAC | 3.03 (0.734) | 3.44 (0.447) | 3.08 (0.685) | 2.83 (0.612)

2. Primary Outcome: Ocular Itching at Day 6
Description: Post-CAC ocular itching from Day 0 will be compared to post-CAC ocular itching, post-instillation, on Day 6. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Per Protocol Population (PP)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 8 | 8 | 9
units on a scale
  3 minutes post-CAC | 2.17 (0.781) | 2.19 (1.108) | 2.06 (0.904) | 2.33 (0.76)
  5 minutes post-CAC | 2.44 (0.778) | 2.59 (0.954) | 2.41 (0.963) | 2.53 (0.824)
  7 minutes post-CAC | 2.17 (0.968) | 2.72 (0.891) | 2.31 (1.007) | 2.14 (0.674)

3. Primary Outcome: Ocular Itching at Day 7
Description: Post-CAC ocular itching from Day 0 will be compared to post-CAC ocular itching, post-instillation, on Day 7. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Per Protocol Population (PP)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 8 | 8 | 9
units on a scale
  3 minutes post-CAC | 2.11 (0.858) | 2.28 (1.004) | 2.09 (1.069) | 2.03 (1.064)
  5 minutes post-CAC | 2.11 (0.894) | 2.69 (1.007) | 2.03 (0.85) | 1.94 (1.108)
  7 minutes post-CAC | 1.97 (0.956) | 2.75 (0.896) | 1.88 (0.982) | 1.72 (0.93)

4. Primary Outcome: Ocular Itching at Day 27
Description: Post-CAC ocular itching from Day 0 will be compared to post-CAC ocular itching, post-instillation, on Day 27. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Per Protocol Population (PP)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 8 | 8 | 8
units on a scale
  3 minutes post-CAC | 2.14 (1.119) | 2.43 (1.231) | 1.75 (1.433) | 2.03 (0.871)
  5 minutes post-CAC | 2.17 (1.281) | 2.64 (1.189) | 2.09 (1.239) | 1.84 (0.801)
  7 minutes post-CAC | 2.03 (1.314) | 2.64 (1.189) | 2 (1.382) | 1.72 (0.807)

5. Primary Outcome: Ocular Itching at Day 28
Description: Post-CAC ocular itching from Day 0 will be compared to post-CAC ocular itching, post-instillation, on Day 28. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 7 | 8 | 8
units on a scale
  3 minutes post-CAC | 1.83 (1.111) | 2.25 (1.267) | 2.03 (1.404) | 1.75 (0.835)
  5 minutes post-CAC | 1.97 (1.343) | 2.64 (1.24) | 2 (1.482) | 1.78 (0.901)
  7 minutes post-CAC | 1.89 (1.426) | 2.71 (1.228) | 1.78 (1.417) | 1.56 (0.853)

6. Primary Outcome: Ocular Redness at Baseline (Day 0)
Description: A baseline CAC was performed on Day 0. Post-CAC ocular redness from Day 0 will be compared to post-CAC ocular redness, post-instillation, on Day 6, Day 7, Day 27 and Day 28. Ocular redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 9 | 9 | 9
units on a scale
  7 minutes post-CAC | 2.11 (0.651) | 2.11 (0.532) | 1.86 (0.333) | 2.08 (0.354)
  15 minutes post-CAC | 2.33 (0.573) | 2.31 (0.349) | 2.11 (0.182) | 2.25 (0.415)
  20 minutes post-CAC | 2.22 (0.537) | 2.28 (0.384) | 2 (0.125) | 2.06 (0.41)

7. Primary Outcome: Ocular Redness at Day 6
Description: Post-CAC ocular redness from Day 0 will be compared to post-CAC ocular redness, post-instillation, on Day 6. Ocular redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per Protocol Population (PP)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 8 | 8 | 9
units on a scale
  7 minutes post-CAC | 2 (0.515) | 2.22 (0.508) | 1.84 (0.823) | 2.11 (0.858)
  15 minutes post-CAC | 1.97 (0.775) | 2.41 (0.626) | 2.13 (0.327) | 2.28 (0.996)
  20 minutes post-CAC | 2 (0.866) | 2.31 (0.691) | 2.03 (0.452) | 2.17 (0.992)

8. Primary Outcome: Ocular Redness at Day 7
Description: Post-CAC ocular redness from Day 0 will be compared to post-CAC ocular redness, post-instillation, on Day 7. Ocular redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per Protocol Population (PP)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 8 | 8 | 9
units on a scale
  7 minutes post-CAC | 2.08 (0.451) | 1.53 (0.761) | 1.59 (0.706) | 1.59 (0.778)
  15 minutes post-CAC | 1.83 (0.791) | 1.69 (0.894) | 1.59 (0.706) | 1.66 (0.981)
  20 minutes post-CAC | 1.72 (0.765) | 1.78 (0.986) | 1.47 (0.737) | 1.5 (0.973)

9. Primary Outcome: Ocular Redness at Day 27
Description: Post-CAC ocular redness from Day 0 will be compared to post-CAC ocular redness, post-instillation, on Day 27. Ocular redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 7 | 8 | 8
units on a scale
  7 minutes post-CAC | 1.72 (0.701) | 2.14 (0.349) | 1.44 (0.32) | 1.56 (0.776)
  15 minutes post-CAC | 1.72 (0.723) | 2.11 (0.476) | 1.63 (0.567) | 1.72 (0.674)
  20 minutes post-CAC | 1.53 (0.814) | 1.89 (0.575) | 1.53 (0.558) | 1.72 (0.749)

10. Primary Outcome: Ocular Redness at Day 28
Description: Post-CAC ocular redness from Day 0 will be compared to post-CAC ocular redness, post-instillation, on Day 28. Ocular redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
Number analyzed (Participants) | 9 | 7 | 8 | 8
units on a scale
  7 minutes post-CAC | 1.58 (0.82) | 1.96 (0.393) | 1.69 (0.637) | 1.81 (0.788)
  15 minutes post-CAC | 1.81 (0.827) | 2.11 (0.378) | 1.69 (0.753) | 1.94 (0.863)
  20 minutes post-CAC | 1.5 (0.791) | 1.86 (0.476) | 1.69 (0.717) | 1.72 (0.761)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through study completion, approximately one month. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited or observed.
Groups:
- Pred Forte; Pred Mild; Alrex; Tears Naturale: 1 drop in each eye up to 4 times daily during a 4 week period
Arm/Group | Pred Forte | Pred Mild | Alrex | Tears Naturale
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 4/9 | 0/9 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pred Forte (N=9) | Pred Mild (N=9) | Alrex (N=9) | Tears Naturale (N=9)
Stinging upon instillation of dose 1 QD (Morning dose every day) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increase in IOP (5 unit) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste Perversion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning upon instillation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower lid swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Itching secondary to Posion Ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Worsening of Rhinitis 1 hour after instillation of Dose 1 (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening of Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular fatigue sensation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Taste perversion upon instillation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes